CLINICAL TRIAL: NCT03023202
Title: UWCCC Precision Medicine Molecular Tumor Board Registry
Brief Title: UWCCC Molecular Tumor Board Registry
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: UW15068; P30CA014520 (NIH); 1R37CA226526-01A1 (NIH); NCI-2019-06343 (Registry Identifier: NCI Trial ID); 2015-1370 (Other: Institutional Review Board); A533400 (Other: UW Madison); SMPH\UWCCC\GENERAL (Other: UW Madison); Protocol Version 3/24/24 (Other: UW Madison)
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Hematologic Neoplasms; Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects will be asked to give one blood sample and up to two tissue samples (one at diagnossi & one at progression of treatment, which are both standard clinical procedures).
  * Drawing 8 tsp of blood at the first clinic visit, DNA extraction from this blood, additional testing on this blood.
  * Retention of residual tumor tissue for future research.
  * Collection of residual fresh tumor tissue [that was biopsied for clinical reasons], and performing of genetic analyses/retention for future research.
  * Banking of data, blood, and biopsy tissue for future research.
  * Distribution of banked data/blood/biopsied tissue for research projects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PMMTB: This study of the PMMTB will include all patients >= 18 with clinically suspected or histologically confirmed solid or hematological malignancy who will undergo genetic testing of their tumor.
  All standard of care functions will be performed by standard procedures.
  Interventions: Other: PMMTB (Precision Medicine Molecular Tumor Board)

INTERVENTIONS:
Other: PMMTB (Precision Medicine Molecular Tumor Board) — PMMTB is a clinical intervention, NOT a research intervention. The research component of this study is to observe the outcomes of the PMMTB.

SUMMARY:
This study seeks to evaluate the clinical utility of the Precision Medicine Molecular Tumor Board, and to track patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinically suspected or histologically confirmed solid or hematological malignancy
* Undergoing genetic testing of tumor
* Ability to understand written informed consent document
* Willingness to sign written informed consent document

Exclusion Criteria:

* Pediatric patients (age<18 years) will be excluded due to a lack of expertise on the molecular tumor committee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include all patients age ≥18 with clinically suspected or histologically confirmed solid or hematological malignancy who will undergo genetic testing of their tumor. It will require each patient to have the ability to understand and willingness to sign a written informed consent document.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-03-30 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Frequency of acceptance of molecular tumor board recommendations | Up to 5 years
  How often the molecular tumor board's recommendations are accepted
Benefit from PMMTB recommended treatment | Up to 5 years
  Whether patients benefit from PMMTB recommended treatment

SECONDARY OUTCOMES:
Correlation of mutations with protein overexpression | Up to 5 years
  Correlate mutations identified in tumor tissue with protein overexpression
Correlations of mutations with circulating tumor DNA | Up to 5 years
  Correlate mutations identified in tumor tissue with circulating tumor DNA
Correlations of mutations with spheroid culture investigations | Up to 5 years
  Correlate mutations identified in tumor tissue with spheroid culture investigations

CONTACTS AND LOCATIONS:
Overall Officials: Mark Burkard, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UW Carbone Cancer Center Home Page — https://cancer.wisc.edu/